CLINICAL TRIAL: NCT04680481
Title: Traveling Wave Transcranial Alternating Current Stimulation for the Control of Large-Scale Brain Networks
Brief Title: Non-Invasive Brain Stimulation to Control Large-Scale Brain Networks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: STUDY00004009; RF1MH124909 (NIH)
Record Dates: First submitted 2020-12-14; First posted 2020-12-23 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Working Memory
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Stimulation Theta Group (Experimental): Participants will experience traveling wave transcranial alternating current stimulation over the fronto-parietal regions at 4 Hz (theta condition).
  Interventions: Device: Transcranial alternating current stimulation
- Stimulation Beta Group (Experimental): Participants will experience traveling wave transcranial alternating current stimulation over the fronto-parietal regions at 23 Hz (beta condition).
  Interventions: Device: Transcranial alternating current stimulation

INTERVENTIONS:
Device: Transcranial alternating current stimulation — Traveling wave transcranial alternating current stimulation will be applied at 4 Hz and 23 Hz over frontal and parietal brain areas in a randomized counterbalanced order.

SUMMARY:
This project will assess the feasibility of traveling wave transcranial alternating current stimulation (tACS) to modify working memory performance and large-scale brain connectivity in surgical epilepsy patients.

ELIGIBILITY:
Inclusion Criteria:

1. the patient can consent for themselves;
2. the patient has or is scheduled for surgically implanted electrodes for the purposes of phase II epilepsy surgical evaluation;
3. age 18+ years old;

Exclusion Criteria:

1. diminished capacity to consent;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Electrophysiological outcomes | Immediate effect during stimulation
  Changes in spectral power and coherence of the local field potentials during transcranial electric stimulation relative to no stimulation periods.
Working memory outcomes | Immediate effect during stimulation
  Changes in working memory performance as measured with the N-back task (quantified with d-prime) during stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Opitz, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared following the IRB guidelines and Data Sharing Policy for the National Institute of Mental Health (NOT-MH-19-033).